CLINICAL TRIAL: NCT01139866
Title: A Multi-Center, Prospective, Observational, Extension Trial Following DURECT Protocol C803-017 to Investigate the Long-term Safety of SABER™-Bupivacaine Following Arthroscopic Shoulder Surgery
Brief Title: An Extension Trial to Evaluate Long-term Safety of SABER™-Bupivacaine for Pain Following Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Durect (Industry)
Collaborators: Nycomed (Industry); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C803-017e
Record Dates: First submitted 2010-05-25; First posted 2010-06-09 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pain
Keywords: Long-term Safety; Shoulder Surgery; bupivacaine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: SABER™-Bupivacaine: Received 5.0 mL SABER™-Bupivacaine in previous C803-017 trial
- Group 2: SABER™-Placebo: Received 5.0 mL SABER™-Placebo in previous C803-017 trial

SUMMARY:
This is an extension to a previous research trial testing SABER™-Bupivacaine (an experimental pain-relieving medication). The purpose of this extension trial is to assess whether treatment with SABER™-Bupivacaine or SABER™-Placebo has had any effect on healing of the participant's shoulder, wound, or the skin near their scar. This trial will also assess safety (side effects).

DETAILED DESCRIPTION:
This research trial will involve all available subjects who received treatment in DURECT Protocol C803-017. All subjects will have the same follow-up safety assessments performed. No experimental treatment will be given in this trial. Subjects, Investigators, and caregivers will remain blinded to the treatment subjects received in the previous trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have provided written consent to participate in the trial prior to any trial procedures and understand that they are free to withdraw from the trial at any time.
* Participants must be able to read and understand the consent form, complete trial-related procedures, and communicate with the trial staff.
* Participants must have participated in DURECT Protocol C803-017 and received SABER™-Bupivacaine or SABER™-Placebo approximately 18 months before enrolling in this trial.

Exclusion Criteria:

* Participants who participated in any other trial with an investigational drug or device since their participation in DURECT protocol C803-017.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All available subjects who received treatment in DURECT protocol C803-017.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety Summaries: Pain Intensity on Movement Evaluation; Surgical Site Healing and Local Tissue Evaluation; Shoulder Examination; MRI; Medical History Update; Adverse Events; and Concomitant Medications | 18 months post-dose in C803-017 trial

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, MD, Study Director — Durect
Locations (8):
- Australia (6):
  - Westmead, New South Wales
  - Auchenflower, Queensland
  - Adelaide, South Australia
  - Toorak Gardens, South Australia
  - Geelong, Victoria
  - Ringwood East, Victoria
- New Zealand (2):
  - Christchurch
  - Hamilton